CLINICAL TRIAL: NCT05199649
Title: Correlation Between the Efficacy of Neoadjuvant Chemotherapy Combined With Immunotherapy of Operable Thoracic Esophageal Squamous Cell Carcinoma and the Metabolites of Intestinal Flora
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20211211
Record Dates: First submitted 2021-12-13; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-12

CONDITIONS: Esophageal Squamous Cell Carcinoma; Intestinal Flora
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm Sintilimab (Experimental): Sintilimab Combined With Chemotherapy
  Interventions: Drug: SintilimabCombined With Chemotherapy

INTERVENTIONS:
Drug: SintilimabCombined With Chemotherapy — Sintilimab and chemotherapy are carried out at the same time for every 3 weeks

SUMMARY:
This study collects stool, blood, and tumor tissue samples from patients with locally advanced esophageal cancer after receiving Sintilimab and chemotherapy to explore the efficacy and intestinal microbes of chemotherapy combined with neoadjuvant immunotherapy for locally advanced operable thoracic esophageal squamous cell carcinoma The main purpose is the relationship between its metabolites, and it will also explore the changes of intestinal flora diversity and metabolites before and after esophageal squamous cell carcinoma chemotherapy combined with immune neoadjuvant therapy

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old and ≤75 years old; 2) Patients with stage I~III thoracic esophageal squamous cell carcinoma diagnosed by histopathological examination (excluding mixed adenosquamous carcinoma and other pathological types); 3) ECOG PS score is 0 or 1; 4) It has sufficient organ and bone marrow function.

Exclusion Criteria:

1. Refuse to participate;
2. Patients who have a higher risk of bleeding or perforation due to the tumor's obvious invasion of the adjacent organs (aorta or trachea) of the esophageal lesion, or patients who have formed a fistula;
3. Have previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibody therapy, or any other antibodies targeting T cell costimulation or checkpoint pathways as specific targets or drug;
4. Participate in another interventional clinical study at the same time, unless participating in an observational (non-interventional) clinical study or in the follow-up phase of an interventional study;
5. Have received systemic systemic treatment with anti-tumor indications Chinese herbal medicine or immunomodulatory drugs (including thymosin, interferon, interleukin, etc.) within 2 weeks before the first administration;
6. Have used immunosuppressive drugs within 1 week before enrollment, excluding nasal spray, inhalation or other local glucocorticoids or physiological doses of systemic glucocorticoids (ie no more than 10mg/day prednisone Or equivalent doses of other glucocorticoids), or use hormones to prevent allergy to contrast agents.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Species and abundance of gut microbiota | 2 year
  Alpha-diversity of samples, that measures both the richness and diversity of species within a group, was calculated on taxa that were observed at least once.
  Beta-diversity, that measures the differences in microbiome composition between groups.

SECONDARY OUTCOMES:
Explore the changes of intestinal flora and metabolomics before and after medication | 2 year
  Discovery of gut microbes and metabolic markers that can predict the efficacy of chemotherapy combined with neoadjuvant immunotherapy for esophageal squamous cell carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of soochow university, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lavelle A, Sokol H. Gut microbiota-derived metabolites as key actors in inflammatory bowel disease. Nat Rev Gastroenterol Hepatol. 2020 Apr;17(4):223-237. doi: 10.1038/s41575-019-0258-z. Epub 2020 Feb 19. PMID 32076145
- [Result] Wilson AJ, Chueh AC, Togel L, Corner GA, Ahmed N, Goel S, Byun DS, Nasser S, Houston MA, Jhawer M, Smartt HJ, Murray LB, Nicholas C, Heerdt BG, Arango D, Augenlicht LH, Mariadason JM. Apoptotic sensitivity of colon cancer cells to histone deacetylase inhibitors is mediated by an Sp1/Sp3-activated transcriptional program involving immediate-early gene induction. Cancer Res. 2010 Jan 15;70(2):609-20. doi: 10.1158/0008-5472.CAN-09-2327. Epub 2010 Jan 12. PMID 20068171
- [Result] Mager LF, Burkhard R, Pett N, Cooke NCA, Brown K, Ramay H, Paik S, Stagg J, Groves RA, Gallo M, Lewis IA, Geuking MB, McCoy KD. Microbiome-derived inosine modulates response to checkpoint inhibitor immunotherapy. Science. 2020 Sep 18;369(6510):1481-1489. doi: 10.1126/science.abc3421. Epub 2020 Aug 13. PMID 32792462
- [Result] Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol. 2021 Jan;19(1):55-71. doi: 10.1038/s41579-020-0433-9. Epub 2020 Sep 4. PMID 32887946
- [Result] Ocvirk S, Wilson AS, Posma JM, Li JV, Koller KR, Day GM, Flanagan CA, Otto JE, Sacco PE, Sacco FD, Sapp FR, Wilson AS, Newton K, Brouard F, DeLany JP, Behnning M, Appolonia CN, Soni D, Bhatti F, Methe B, Fitch A, Morris A, Gaskins HR, Kinross J, Nicholson JK, Thomas TK, O'Keefe SJD. A prospective cohort analysis of gut microbial co-metabolism in Alaska Native and rural African people at high and low risk of colorectal cancer. Am J Clin Nutr. 2020 Feb 1;111(2):406-419. doi: 10.1093/ajcn/nqz301. PMID 31851298